CLINICAL TRIAL: NCT00935168
Title: A Multi-centre Randomized Controlled Trial of Fluid Resuscitation With Starch (6%Hydroxyethyl Starch 130/0.4) Compared to Saline (0.9% Sodium Chloride) in Intensive Care Patients on Mortality
Brief Title: Crystalloid Versus Hydroxyethyl Starch Trials
Acronym: CHEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Sydney (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network); Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI-CCT24378; ACTRN12609000245291 (Registry Identifier: Australian and New Zealand Clinical Trial Registry)
Record Dates: First submitted 2009-07-01; First posted 2009-07-08 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-02

CONDITIONS: Intensive Care
Keywords: Intensive Care; Fluid Resuscitation; Saline; Hydroxy-ethyl starch
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxy-ethyl starch (Experimental): Intravenous fluid resuscitation with 6% Hydroxy-ethyl starch (130/0.4)
  Interventions: Drug: 6% Hydroxy-ethyl starch (130/0.4)
- Saline (Active Comparator): Intravenous fluid resuscitation with saline (0.9% sodium chloride)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: 6% Hydroxy-ethyl starch (130/0.4) — Maximum dose of 50ml/kg/day of 6% hydroxy-ethyl starch (130/0.4) for intravascular volume fluid resuscitation
  Other Names: Voluven 6%
  Arms: Hydroxy-ethyl starch
Drug: Saline — Maximum dose of 50ml/kg/day of saline for intravascular volume fluid resuscitation
  Other Names: Sodium Chloride 0.9%
  Arms: Saline

SUMMARY:
The aim of this study is to determine whether patients in the Intensive Care Unit who receive fluid resuscitation with either hydroxyethyl starch (a synthetic colloid solution) or saline (a salt solution), have an increased rate of survival at 90 days.

DETAILED DESCRIPTION:
Patients in intensive care units frequently require intravenous fluid because the treating clinicians consider that the patient's blood pressure or circulating blood volume needs to be increased to clinically acceptable levels. Despite fluid resuscitation being a fundamental part of standard medical treatment for critically ill patients, clinicians are left with uncertainty about the optimal choice and volume of fluid that should be administered.

This study is a prospective, multi-centre, blinded, randomised controlled trial.

The two fluids being compared are 0.9% sodium chloride (saline) and 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride,(starch). The null hypothesis assumes no difference in all-cause mortality between patients given starch in comparison with patients given saline for fluid resuscitation.

Each patient who meets all inclusion criteria and none of the exclusion criteria will be randomised to receive one of the two study fluids for fluid resuscitation.

Once treatment has been assigned the participant will continue to receive either starch or saline only for all fluid resuscitation requirements in intensive care. The treating clinical team will decide the amount and frequency of the fluid given for resuscitation based on standard care.

During their ICU stay, participants will have information on the use of study fluids, other fluids, kidney function, blood pressure, heart rate and other haemodynamic data that is routinely recorded in the medical record collected. All participants will be followed up at day 90 and at 6 months after randomisation.

The participants status (alive, in hospital and length of stay) will be recorded at day 28 and day 90 after randomisation. At the 6 month follow-up all participants or their carer will be interviewed by telephone using standardised questionnaires about the participant's quality of life. In addition, participants who were admitted to intensive care with a traumatic brain injury will be interviewed to determine how well the participant is recovering.

After all patients have completed the 6 months of follow-up, data linkage will also be used to link patients (in NSW only) to health databases in order to obtain information on their use of health services.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained or if not possible, the procedure for obtaining informed consent has been approved by the ethics committee.
* Fluid resuscitation is required to increase or maintain intravascular volume that is in addition to maintenance fluids, enteral and parenteral nutrition, blood products and specific replacement fluids to replace ongoing insensible or fluid losses from other sites (e.g., fistula losses from the gastrointestinal tract, urinary losses from diabetes insipidus or the polyuric phase of acute renal failure or to correct metabolic derangements).
* The ICU clinician considers that both 6% hydroxyethyl starch (130/0.4) and saline are equally appropriate for the patient and that no specific indication or contraindication for either exists.
* The requirement for fluid resuscitation must be supported by AT LEAST ONE of the following clinical signs:

  1. Heart rate > 90 beats per minute
  2. Systolic blood pressure (SBP) < 100mmHg or mean arterial pressure (MAP) < 75mmHg or at least 40mmHg decrease in SBP or MAP from the baseline recording
  3. Central venous pressure < 10mmHg
  4. Pulmonary artery wedge pressure < 12 mmHg
  5. Respiratory variation in systolic or mean arterial blood pressure of >5 mmHg
  6. Capillary refill time > one second
  7. Urine output < 0.5 ml/kg for one hour

Exclusion Criteria:

* Previous allergic reaction to hydroxyethyl starch solution.
* Primary non-traumatic intracranial haemorrhage or severe traumatic intracranial haemorrhage (mass lesion > 25 ml).
* Patients who are receiving renal replacement therapy or in whom the ICU physician considers renal replacement therapy is imminent (i.e. renal replacement therapy will start in 6 hours)
* Patients with documented serum creatinine value ≥ 350µmol/L and urine output averaging ≤ 10ml / hr over 12 hours
* Severe hypernatraemia (Serum sodium > 160 mmol/l) or severe hyperchloraemia (Serum chloride > 130 mmol/l).
* Women of child bearing age (18-49 years old), unless evidence of documented menopause, hysterectomy or surgical sterilisation or negative pregnancy test before randomisation
* Breastfeeding
* Patients who have received > 1000mL hydroxyethyl starch in the 24 hours before randomization.
* Patients admitted to the ICU following cardiac surgery; patients admitted to ICU following cardiac surgery.
* Patients admitted to the ICU for the treatment of burns or following liver transplantation surgery.
* Death is deemed imminent and inevitable or the patient has an underlying disease process with a life expectancy of < 90 days.
* A limitation of therapy order has been documented restricting implementation of the study protocol or the treating clinician deems aggressive care unsuitable.
* Patient has previously been enrolled in the CHEST study.
* Patient has previously received fluid resuscitation that was prescribed within the study ICU during this current ICU admission.
* Patient has been transferred to the study ICU from another ICU and received fluid resuscitation for the treatment of volume depletion in that other ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 90 days

SECONDARY OUTCOMES:
Renal failure requiring renal replacement therapy will be assessed using hospital records. | During intensive care Unit (ICU) stay after randomisation up to 90 days
Other organ failures will be assessed using the Sequential Organ Failure Assessment (SOFA) score which is based on biochemical and bio-physiological parameters recorded in the hospital record. | During ICU stay after randomisation up to 90 days
ICU, hospital and 28 day mortality | At 28 days and 6 months after randomisation
Quality of life will be assessed using the EQ-5D questionnaire. | 6 months after randomisation
Functional status will be assessed using the Glasgow Outcome score. | 6 months after randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: John A Myburgh, PhD FJFICM, Study Chair — The George Institute; Simon Finfer, Principal Investigator — Royal North Shore Hospital, NSW, Australia; David Gattas, Principal Investigator — Royal Prince Alfred Hospital, NSW, Australia; Eddie Stachowski, Principal Investigator — Westmead Hospital, NSW, Australia; Michael Parr, Principal Investigator — Liverpool Hospital, NSW, Australia; Ian Seppelt, Principal Investigator — Nepean Hospital, NSW, Australia; Peter Harrigan, Principal Investigator — John Hunter Hospital, NSW, Australia; Rinaldo Bellomo, Principal Investigator — Austin Hospital, VIC, Australia; Forbes McGain, Principal Investigator — Western Hospital, VIC, Australia; Rob Boots, Principal Investigator — Royal Brisbane & Women's Hospital, QLD, Australia; Jason Fletcher, Principal Investigator — Bendigo Health, VIC, Australia; David Milliss, Principal Investigator — Concord Hospital, NSW, Australia; Benno Ihle, Principal Investigator — Epworth Richmond, VIC, Australia; David Ernest, Principal Investigator — Box Hill Hospital, VIC, Australia; Jeffrey Presneill, Principal Investigator — Mater Health Services, QLD, Australia; Claire Cattigan, Principal Investigator — Geelong Hospital, VIC, Australia; Katrina Ellem, Principal Investigator — Calvary Mater Newcastle, NSW, Australia; Seton Henderson, Principal Investigator — Christchurch Hospital, New Zealand; Shay McGuinness, Principal Investigator — Auckland CVICU, New Zealand; Dick Dinsdale, Principal Investigator — Wellington Hospital, New Zealand; Michael Reade, Principal Investigator — The Northen Hospital, VIC, Australia; Bart de Keulenaer, Principal Investigator — Fremantle Hospital, WA, Australia; Latesh Poojara, Principal Investigator — Blacktown Hospital, NSW, Australia; Yahya Shehabi, Principal Investigator — Prince of Wales Hospital, NSW, Australia; Imogen Mitchell, Principal Investigator — The Canberra Hospital, ACT, Australia; John Santamaria, Principal Investigator — St Vincent's Hospital, VIC, Australia; Troy Browne, Principal Investigator — Tauranga Hospital, New Zealand; Kavi Haji, Principal Investigator — Frankston Hospital, VIC Australia; Frank van Haren, Principal Investigator — Waikato Hospital, New Zealand; Janet Liang, Principal Investigator — North Shore Hospital, New Zealand; Bala Venkatesh, Principal Investigator — Wesley Hospital, VIC, Australia; David Cooper, Principal Investigator — Royal Hobart Hospital, TAS, Australia; John Myburgh, Principal Investigator — St George Hospital, NSW, Australia
Locations (1):
- The George Institute for International Health, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Taylor C, Thompson K, Finfer S, Higgins A, Jan S, Li Q, Liu B, Myburgh J; Crystalloid versus Hydroxyethyl Starch Trial (CHEST) investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Hydroxyethyl starch versus saline for resuscitation of patients in intensive care: long-term outcomes and cost-effectiveness analysis of a cohort from CHEST. Lancet Respir Med. 2016 Oct;4(10):818-825. doi: 10.1016/S2213-2600(16)30120-5. Epub 2016 Jun 17. PMID 27324967
- [Derived] Phillips DP, Kaynar AM, Kellum JA, Gomez H. Crystalloids vs. colloids: KO at the twelfth round? Crit Care. 2013 May 29;17(3):319. doi: 10.1186/cc12708. PMID 23731998
- [Derived] Myburgh JA, Finfer S, Bellomo R, Billot L, Cass A, Gattas D, Glass P, Lipman J, Liu B, McArthur C, McGuinness S, Rajbhandari D, Taylor CB, Webb SA; CHEST Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Hydroxyethyl starch or saline for fluid resuscitation in intensive care. N Engl J Med. 2012 Nov 15;367(20):1901-11. doi: 10.1056/NEJMoa1209759. Epub 2012 Oct 17. PMID 23075127